CLINICAL TRIAL: NCT00432900
Title: PET Evaluation of Brain Peripheral Benzodiazepine Receptors Using [(11)C]PBR28 in Patients With Multiple Sclerosis (MS)
Brief Title: Brain Peripheral Benzodiazepine Receptors in Patients With Multiple Sclerosis
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 070092; 07-N-0092
Record Dates: First submitted 2007-02-07; First posted 2007-02-08 (Estimated); Last update posted 2019-12-12 (Actual); Status verified 2014-04-22

CONDITIONS: Multiple Sclerosis
Keywords: Inflammation; Neuroimmunology; Multiple Sclerosis; MS; Healthy Volunteer; HV
MeSH Terms: conditions — Multiple Sclerosis; Inflammation

ARMS (2):
- Healthy Volunteer (Active Comparator): Healthy Volunteers
  Interventions: Radiation: [(11)C]PBR28
- Patient (Experimental): Multiple Sclerosis Patients
  Interventions: Radiation: [(11)C]PBR28

INTERVENTIONS:
Radiation: [(11)C]PBR28 — PET Ligand

SUMMARY:
This study will use positron emission tomography (PET) to measure a brain protein called peripheral benzodiazepine receptor (PBR) in patients with multiple sclerosis. PBR is created during the inflammation process, and brain inflammation is a key feature of multiple sclerosis (MS). PBR usually affects one type of brain cell, but it can also cause damage to surrounding areas of the brain in patients with MS. PET studies of PBRs and brain inflammation may help elucidate the role of these brain cells in patients with MS.

Healthy normal volunteers and patients with MS between 18 and 70 years of age may be eligible for this study. Patients with MS must have had onset of disease between 18 and 40 years of age.

Patients with MS undergo the following procedures:

Visit 1: Medical history, physical examination, blood tests and magnetic resonance imaging (MRI).

Visit 2: Blood tests and PET scan.

Visits 3 and 4: MRI and physical examination.

Visit 5: PET scan and blood tests.

Visit 6: MRI and physical examination.

Healthy volunteers undergo the following:

Visit 1: Medical history, physical examination, blood tests.

Visits 2 and 3: PET and blood tests.

Magnetic Resonance Imaging

MRI uses a magnetic field and radio waves to produce images of body tissues and organs. For this procedure, the subject lies on a table that can slide in and out of the scanner (a metal cylinder), wearing earplugs to muffle loud knocking noises that occur during the scanning process. The procedure lasts about 90 minutes; the patient is asked to lie still for up to 25 minutes at a time. The subject can communicate with the MRI staff at all times during the scan. During part of the scan a contrast agent is administered through a catheter (plastic tube) placed in an arm vein to enhance the images.

Positron Emission Tomography (PET)

The PET scan gives information on brain and body chemistry and function. The subject lies on a bed that slides in and out of the doughnut-shaped scanner. A catheter is placed in a vein in the arm and another is placed in an artery in the wrist or elbow area. The catheter in the arm is used for injecting a radioactive material that the scanner detects, and the other is used to collect blood samples. A custom-molded plastic mask is used to support the head and prevent it from moving during the procedure. The subject may be asked to perform various tasks during the PET scan or to lie quietly. The scan lasts about 2.5 hours.

DETAILED DESCRIPTION:
OBJECTIVE:

The primary objective of this study is to measure brain peripheral benzodiazepine receptor (PBR) expression as a marker of neuroinflammation in subjects with MS using [(11)C]PBR28 PET imaging. Inflammation in the central nervous system (CNS) is a prominent feature of multiple sclerosis (MS), the leading cause of neurological disability in young adults. A complex sequence of inflammatory events leads to the formation of new lesions. The disruption of blood-brain barrier that occurs during this inflammatory cascade is the basis of Gadolinium-DTPA (Gd-DTPA) enhancing lesion on magnetic resonance imaging (MRI), currently the most widely utilized marker of neuroinflammation in MS. Although Gd-DTPA enhancement correlates with acute clinical relapses, its limitation as a biomarker of disease activity includes the relative insensitivity to mild degrees of inflammation and the lack of correlation to long-term disability. An alternative marker of neuroinflammation may, therefore, be informative. Activated microglia and macrophage constitute the secondary effector cells of CNS inflammation in MS. Recent studies investigating the expression of the peripheral benzodiazepine receptor (PBR) in the CNS have shown that the increased expression of PBR is a marker of activated microglia/macrophage. Specific ligands for PBR have allowed the study of activated microglia/macrophage in vivo through positron emission tomography (PET) imaging in a number of settings including inflammatory, ischemic and toxic injury to the CNS. The availability of a novel PBR ligand [(11)C]PBR28 developed by the Molecular Imaging Branch, NIMH, that demonstrated greater specific signal for PBR than the previously available ligands affords a unique opportunity to investigate a cell-type specific marker of neuroinflammation in MS.

STUDY POPULATION:

Subjects with definite MS (McDonald criteria) with evidence of brain inflammatory activity indicated by presence of Gd-DTPA enhancing lesions on MRI and a control group consisting of age-matched healthy volunteers.

DESIGN:

Up to 32 subjects with MS will undergo screening TSPO genotype analysis by PCR to accrue up to 16 MS subjects with confirmed high- or mixed- affinity binding genotype (HL or HH genotype) who will undergo a brain [(11)C]PBR28 PET and MRI imaging. Subjects with MS will undergo follow-up brain [(11)C]PBR28 PET and MRI at approximately 4-month interval. Subjects will undergo clinical examination at each PET imaging time point to assess clinical measures of disability and impairment. Up to an equal number of age-matched healthy volunteers will undergo screening TSPO genotype analysis by PCR. Up to 16 healthy volunteers with confirmed high- or mixed- affinity binding genotype (HL or HH genotype)undergo test retest brain [(11)C]PBR28 PET studies to determine the reproducibility of [(11)C]PBR28 PET in a healthy population compared to MS.

OUTCOME MEASURES:

The study seeks to test PBR expression measured by [(11)C]PBR28 PET imaging as a marker of neuroinflammation in patients with MS. Primary outcome measures include 1) correlation between increased PBR expression and gadolinium-enhancing lesions on MRI, and 2) correlation between increased PBR expression and previously and/or persistently gadolinium-enhancing lesions on MRI, 3) PBR expression in subjects with multiple sclerosis compared to that in healthy volunteers.

ELIGIBILITY:
* SUBJECTS WITH MULTIPLE SCLEROSIS - INCLUSION CRITERIA:
* Ages between 18 and 70, inclusive.
* Diagnosis of definite MS according to published criteria.
* The presence of at least one gadolinium-enhancing lesion on the screening brain magnetic resonance image (MRI), and T2 lesion load volume greater than 5 cc.
* Subjects must be able to provide written, informed consent prior to any testing under this protocol, including screening and baseline investigations that are not considered part of routine patient care.

SUBJECTS WITH MULTIPLE SCLEROSIS - EXCLUSION CRITERIA:

* Prior participation in other research protocols or clinical care in the last year such that radiation exposure would exceed the annual guidelines.
* Homozyous for the low- affinity binding form of TSPO by TSPO genotype analysis ( Ala147Thr polymorphism in rs6971 SNP in exon 4 of the TSPO gene).
* Pregnancy and breast-feeding.
* Presence of ferromagnetic metal in the body or heart pacemaker.
* ECG with clinically significant abnormalities.
* Positive HIV test.
* Positive pregnancy test.
* Concurrent medical conditions including hepatic cirrhosis, end-stage renal disease or any acute and severe decompensation of disease that in the opinion of the investigator would compromise the safety of the patient.
* Subjects with cognitive impairment who are unable to provide written, informed consent.
* Subjects who have received immunomodulatory/disease-modifying therapy, including investigational MS therapy, within 12 weeks prior to PET imaging or who have received corticosteroids within 6 weeks prior to PET imaging.

HEALTHY VOLUNTEERS - INCLUSION CRITERIA:

All subjects must be healthy and aged 18-70 years.

HEALTHY VOLUNTEERS - EXCLUSION CRITERIA:

Homozyous for the low- affinity binding form of TSPO by TSPO genotype analysis ( Ala147Thr polymorphism in rs6971 SNP in exon 4 of the TSPO gene).

Current psychiatric illness, substance abuse or severe systemic disease based on history and physical exam.

ECG with clinically significant abnormalities. Any existing physical exam and ECG within one year will be reviewed and if none already exists in the chart, these will be obtained and reviewed.

Laboratory tests with clinically significant abnormalities.

Prior participation in other research protocols in the last year such that radiation exposure would exceed the annual guidelines.

Pregnancy and breast-feeding.

Positive pregnancy test.

Claustrophobia.

Presence of ferromagnetic metal in the body or heart pacemaker.

Positive HIV test.

A history of brain disease.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2007-02-05; Primary Completion 2013-05-23 (Actual); Study Completion 2013-05-29 (Actual)

PRIMARY OUTCOMES:
Correspondence between increased PBR expression measured by [11C]PBR28 PET and gadolinium-enhancing lesions on MRI. | At time of dosing
Correspondence between increased PBR expression and previously and/or persistently gadolinium-enhancing lesions on MRI. | At time of dosing

SECONDARY OUTCOMES:
Correspondence between PBR expression and other MRI defined pathology including T2-weighted hyperintense and T1-weighted hypointense lesions. | Follow-up (~Month 4)
Correspondence between PBR expression and normal appearing white and gray matter on MRI. | Follow-up (~Month 4)

CONTACTS AND LOCATIONS:
Overall Officials: Steven Jacobson, Ph.D., Principal Investigator — National Institute of Neurological Disorders and Stroke (NINDS)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] McDonald WI, Compston A, Edan G, Goodkin D, Hartung HP, Lublin FD, McFarland HF, Paty DW, Polman CH, Reingold SC, Sandberg-Wollheim M, Sibley W, Thompson A, van den Noort S, Weinshenker BY, Wolinsky JS. Recommended diagnostic criteria for multiple sclerosis: guidelines from the International Panel on the diagnosis of multiple sclerosis. Ann Neurol. 2001 Jul;50(1):121-7. doi: 10.1002/ana.1032. PMID 11456302
- [Background] Noseworthy JH, Lucchinetti C, Rodriguez M, Weinshenker BG. Multiple sclerosis. N Engl J Med. 2000 Sep 28;343(13):938-52. doi: 10.1056/NEJM200009283431307. No abstract available. PMID 11006371
- [Background] Cotton F, Weiner HL, Jolesz FA, Guttmann CR. MRI contrast uptake in new lesions in relapsing-remitting MS followed at weekly intervals. Neurology. 2003 Feb 25;60(4):640-6. doi: 10.1212/01.wnl.0000046587.83503.1e. PMID 12601106